CLINICAL TRIAL: NCT00703716
Title: Stabilization of Trochanteric Fracture Using a Screw-plate TRAUMAX
Acronym: TRAUMAX
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-06
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Hip Fracture
Keywords: mini-invasive; dynamic screw-plate; Surfix; Lock-screw
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the stabilization of trochanteric fracture using a screw-plate TRAUMAX

DETAILED DESCRIPTION:
Hip fractures are a serious public health problem. The current incidence is projected to increase fourfold worldwide by the year 2050. This affliction is obviously linked to the aging of the population and the absence of a systematic prevention of osteoporosis.

This leads to the creation of a minimally invasive, or ever percutaneous, implantable osteosynthesis material which associates :

* the well-known reliability of osteosynthesis using screw-plate with barrel,
* the safety of the fixation with Surfix concept, locking the screws to the plate using lock-screws,
* a modularity thanks to the choice between 3 sizes of barrel,
* the creation of a simple material, easing the operative surgery by minimally invasive approach.

The TRAUMAX answers to all those characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Age > 18
* with a trochanteric fracture whom surgeon advised the use of a screw-plate TRAUMAX

Exclusion Criteria:

* Patient with an acute infection
* Patient with a major osseous deterioration which not allows a correct support of the screws in the bone
* Patient with an ASA score of 4 or 5
* Patient whom the time between the fracture and the surgery could be higher than 8 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a trochanteric fracture whom surgeon advised the use of a screw-plate TRAUMAX
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The consolidation rate | 6 months after surgery
The rate of complication due to the device | 6 months after surgery

SECONDARY OUTCOMES:
The evolution of the functional scores (Parker, ADL, Katz, Robinson) between before the fracture and after the intervention. | 3 and 6 months after surgery
PMA score | 3 and 6 months after surgery
operating time | during the surgery
The duration of the use of the amplifier of brilliancy during the intervention | during the surgery
The radiological position of the device | 5 days, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: CHIRON Philippe, Principal Investigator — CHU Rangueil, Toulouse, FRANCE
Locations (10):
- France (10):
  - Hôpital d'Instruction des Armées R. Picqué, Bordeaux
  - CHU La Cavale Blanche, Brest
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Centre Hospitalier du Nord Mayenne, Mayenne
  - CHU Nantes, Nantes
  - Hopital Saint Antoine, Paris
  - Clinique de l'alliance, Saint-Cyr-sur-Loire
  - Nouvelle Clinique de l'Union et du Vaurais, Saint-Jean
  - CHU Toulouse, Toulouse
  - Centre Hospitalier Saint Cyr, Villeneuve-sur-Lot